CLINICAL TRIAL: NCT02421770
Title: Chamaemelum Nobile 2% Versus Placebo Topic Gel to Treatment Oral LichenPlanus
Brief Title: Chamaemelum Nobile 2% Versus Placebo Topic Gel to Treat Oral Lichen Planus
Acronym: lichenPlanus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, MD, DDS, PhD, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMurcia
Record Dates: First submitted 2015-04-08; First posted 2015-04-21 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Chamaemelum Nobile (Experimental): Experimental Chamaemelum Nobile 2% gel "During the 6-week double-blind phase, all patients will be randomly assigned to receive Chamaemelum Nobile 2% gel twice daily with occlusion on the affected are
  Interventions: Other: Chamaemelum nobile 2%
- Placebo (Placebo Comparator): During the 6-week double-blind phase, all patients will be randomly assigned to receive vehicle ( placebo)twice daily with occlusion on the affected are
  Interventions: Other: placebo

INTERVENTIONS:
Other: Chamaemelum nobile 2% — Experimental Chamaemelum Nobile 2% gel Active "During the 6-week double-blind phase, all patients will be randomly assigned to receive Chamaemelum Nobile 2% gel Active or its vehicle twice daily with occlusion on the affected are
  Arms: Experimental Chamaemelum Nobile
Other: placebo
  Arms: Placebo

SUMMARY:
Oral lichen planus (OLP) is a chronic inflammatory mucocutaneous disease characterized by outbreaks or flares. It affects 0.2-1.9% of the population. Although the etiology is unknown, the pathogenesis of OLP is known to involve an immune disorder, with epithelial damage caused by cytotoxic CD8 + lymphocytes. Clinically, the disease is characterized by different types of lesions - papular, reticular and in the form of plaques - that can alternate with erosive and/or ulcerative areas. A variety of treatments have been proposed for OLP: topical or systemic corticosteroids, cyclosporine, retinoids, azathioprine, tacrolimus, pimecrolimus, photochemotherapy and surgery. Patients with symptomatic OLP often require intensive therapy to reduce the signs and symptoms. The disease can produce considerable morbidity and alter patient quality of life, particularly in the presence of ulcerative lesions.

There is no fully resolutive and effective treatment - the management strategy focusing on the use of drugs that counter tissue inflammation and the underlying immunological mechanisms. The main inconvenience of these treatments is represented by the side effects they usually produce.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate that if Chamaemelum Nobile a can be used in the treatment of oral lichen planus. This could be useful as Chamaemelum Nobile has no reported side effects and hence it can used in place of steroids which are commonly used for this condition and have many reported adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients clinically & histopathologically diagnosed to be suffering from oral lichen planus.
2. Patients who had symptoms i.e. pain and/or burning sensation secondary to oral lichen planus.
3. Patients not on any treatment for the same. In case they were, then such treatment was stopped and a washout period of two weeks was given.

Exclusion Criteria:

1. Patients suffering from any systemic disease/s like
2. Patients with any other mucosal disease or any other skin disease which may be associated with oral lesions.
3. Patients on any drug therapy which may cause lichen planus like lesions.
4. Patients with findings of any physical or mental abnormality, which would interfere with or be affected by the study procedure.
5. Patients with a known allergy or contraindication to study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Relief from signs & symptoms of disease (Visual Analog Scale and change in size of target lesion) | 6 week
  The primary study end-point was the Visual Analog Scale (VAS) score for pain change in the size of the target erosion, erythema at the start and after 6week

CONTACTS AND LOCATIONS:
Overall Officials: Pia Lopez Jornet, MD,DDS,PhD, Principal Investigator — Universidad de Murcia
Locations (1):
- Pia Lopez Jornet, Murcia, Murcia, Spain

REFERENCES:
- [Background] Varoni EM, Lodi G, Sardella A, Carrassi A, Iriti M. Plant polyphenols and oral health: old phytochemicals for new fields. Curr Med Chem. 2012;19(11):1706-20. doi: 10.2174/092986712799945012. PMID 22376030
- [Background] Petti S, Scully C. Polyphenols, oral health and disease: A review. J Dent. 2009 Jun;37(6):413-23. doi: 10.1016/j.jdent.2009.02.003. Epub 2009 Mar 19. PMID 19303186
- [Result] Thongprasom K, Prapinjumrune C, Carrozzo M. Novel therapies for oral lichen planus. J Oral Pathol Med. 2013 Nov;42(10):721-7. doi: 10.1111/jop.12083. Epub 2013 May 13. PMID 23668304
- [Result] Lodi G, Carrozzo M, Furness S, Thongprasom K. Interventions for treating oral lichen planus: a systematic review. Br J Dermatol. 2012 May;166(5):938-47. doi: 10.1111/j.1365-2133.2012.10821.x. Epub 2012 Mar 27. PMID 22242640